CLINICAL TRIAL: NCT06395792
Title: Epidemiology of Dravet and Lennox-Gastaut Syndromes in Portugal
Brief Title: A Study on Dravet Syndrome (DS) and Lennox-Gastaut Syndrome (LGS) in Children, Teenagers and Adults in Portugal
Acronym: DRALEGA-PT
Status: Withdrawn | Type: Observational
Why Stopped: Business Decision
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-935-5004
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Dravet Syndrome (DS); Lennox-Gastaut Syndrome (LGS)
Keywords: Drug Therapy
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With DS or LGS: Participants with a medical record of diagnosis with either DS or LGS that are treated in the participating hospitals and reside in the reference area of these hospitals will be included and data will be retrospectively collected for the period between 01 January 2021 to 31 December 2022.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
The main aim of this study is to learn about the percentage of persons diagnosed with Dravet Syndrome (DS) and Lennox-Gastaut-Syndrome (LGS) in 2022 and of persons newly diagnosed in 2021 and 2022 compared to the overall population in Portugal. Other aims are to understand how many percent of the persons diagnosed with DS and LGS are children, teenagers or adults and gather additional information on diagnosis and persons diagnosed with DS and LGS in Portugal.

Information will be taken from a participant's existing medical hospital records. It is planned to review data in approximately 3 public hospitals in Portugal. No personal information of the participants will be collected.

DETAILED DESCRIPTION:
This is a non-interventional, multicentre, cross-sectional retrospective study of participants from Portugal with Dravet syndrome (DS) and Lennox-Gastaut syndrome (LGS) at public hospitals. The participants will be identified from their medical charts or hospital records and those who meet the eligibility criteria will be included.

This multi-center trial will be conducted in Portugal. Data will be retrospectively collected for the observation period between 01 January 2021 to 31 December 2022. The total duration of the study is approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis criteria for DS:

   • All the following criteria must be met: i. Seizures onset within 1-20 months (usually within the first year of life). ii. Normal initial development prior to presentation (no cognitive or behavioural disability before the onset of seizures) followed by behaviour and cognitive impairment.

   iii. Recurrent focal clonic (hemiclonic) febrile and afebrile seizures (which often alternate sides from seizure to seizure), focal to bilateral tonic-clonic, and/or generalized clonic seizures.

   • And at least one of the following criteria must be met: i. Emergence of other seizure type, including atypical absence seizures, myoclonic seizures, atonic seizures, or non-tonic-clonic status epilepticus between 1-4 years.

   ii. Seizures triggered by fever due to illness or vaccinations, hot baths, sudden temperature changes, high level of activity, or by strong lighting or exposure to certain visual patterns.

   iii. Mutations or copy number variants in the SCN1A gene.
2. Diagnosis criteria for LGS:

Given the uncertainties associated with the diagnosis of this condition, two different criteria will be used, a stricter criterion, intended to identify "pure" Lennox-Gastaut syndrome participants, and a wider criterion, intended to also include the so-called Lennox-Gastaut-like participants.

Lennox-Gastaut syndrome - stricter criteria:

• All the following criteria must be met: i. Seizures onset before 18 years of age, typically from 1 to 8 years. ii. Progressive development/cognition impairment after seizures onset. iii. Tonic seizures. iv. At least one additional seizure: generalised tonic-clonic seizures, atypical absence seizures, atonic seizures, myoclonic seizures, focal impaired awareness, epileptic spams, or non-convulsive status epilepticus v. Slow (less thank [<] 2.5 hertz [Hz]) spike-and-wave EEG pattern. vi. Paroxysmal fast activity (10 Hz or greater) in sleep.

Lennox-Gastaut syndrome - wider criteria:

* At least one the following criteria must be met:

  i. Tonic seizures. ii. Multiple types of seizures, including generalised tonic-clonic seizures, atypical absence seizures, atonic seizures, myoclonic seizures, myoclonic-atonic seizures, focal seizures, epileptic spams, or nonconvulsive status epilepticus.
* And at least one the following criteria must be met:

  i. Slow (<2.5 Hz) spike-and-wave EEG pattern. ii. Paroxysmal fast activity (10 Hz or greater) in sleep.
* And at least two of the following criteria must be met:

  i. Seizures onset before 18 years of age, typically from 1 to 8 years. ii. Progressive development/cognition impairment after seizures onset. iii. Development/cognition impairment starts prior to seizures onset. iv. History of Infantile epileptic spasms syndrome (IESS), West or Ohtahara syndromes.

Exclusion Criteria

1. Has epileptic condition other than DS or LGS.
2. Has DS or LGS not residents in the reference area of the hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with DS or LGS at public hospitals in Portugal will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
One-Year Period Prevalence of DS | Up to 12 months
  Number of participants with DS over a period of one year will be assessed.
Incidence of DS | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Number of participants diagnosed annually with DS yearly.
One-Year Period Prevalence of LGS Based on Stricter Diagnosis Criterion | Up to 12 months
  Number of participants with LGS over a period of one year based on stricter diagnosis criterion will be assessed.
Incidence of LGS Based on Stricter Diagnosis Criterion | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Number of participants diagnosed annually with LGS based on stricter diagnosis criterion.

SECONDARY OUTCOMES:
One-Year Period Prevalence of LGS Based on Wider Diagnosis Criterion | Up to 12 months
  Number of participants with LGS over a period of one year based on wider diagnosis criterion will be assessed.
Incidence of LGS Based on Wider Diagnosis Criterion | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Number of participants diagnosed annually with LGS based on wider diagnosis criterion.
One-Year Period Prevalence of Paediatric DS | Up to 12 months
  Number of participants with paediatric DS over a period of one year will be assessed.
One-Year Period Prevalence of Paediatric LGS Based on Stricter and Wider Diagnoses Criteria | Up to 12 months
  Number of participants with paediatric LGS over a period of one year based on stricter and wider diagnoses criteria will be assessed.
One-Year Period Prevalence of Adult DS | Up to 12 months
  Number of participants with adult DS over a period of one year will be assessed.
One-Year Period Prevalence of Adult LGS Based on Stricter and Wider Diagnoses Criteria | Up to 12 months
  Number of participants with adult LGS over period of one year based on stricter and wider diagnoses criteria will be assessed.
Incidence of Paediatric DS | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Number of paediatric participants diagnosed annually with DS.
Incidence of Paediatric LGS Based on Stricter and Wider Diagnoses Criteria | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Number of paediatric participants diagnosed annually with LGS based on stricter and wider diagnoses criteria.
Incidence of Adult DS | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Number of adult participants diagnosed annually with DS.
Incidence of Adult LGS Based on Stricter and Wider Diagnoses Criteria | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Number of adult participants diagnosed annually with LGS based on stricter and wider diagnoses criteria.
DS Categorized Based on Gender Distribution | Up to 12 months
  DS categorized participants based on gender distribution will be assessed.
LGS Categorized Based on Gender Distribution According to Stricter and Wider Diagnoses Criteria | Up to 12 months
  LGS categorized participants based on gender distribution according to Stricter and Wider diagnoses criteria will be assessed.
DS Categorized Based on Age Distribution | Up to 12 months
  DS categorized participants based on age distribution will be assessed.
LGS Categorized Based on Age Distribution According to Stricter and Wider Diagnoses Criteria | Up to 12 months
  LGS categorized participants based on age distribution according to Stricter and Wider diagnoses criteria will be assessed.
DS Categorized Based on Gender Distribution at Diagnosis | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Annually diagnosed DS participants will be categorized based on gender distribution at diagnosis.
LGS Categorized Based on Gender Distribution at Diagnosis According to Stricter and Wider Diagnoses Criteria | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Annually diagnosed LGS participants will be categorized based on gender distribution at diagnosis.
DS Categorized Based on Age Distribution at Diagnosis | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Annually diagnosed DS participants will be categorized based on age distribution at diagnosis.
LGS Categorized Based on Age Distribution at Diagnosis According to Stricter and Wider Diagnoses Criteria | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Annually diagnosed LGS participants will be categorized based on age distribution at diagnosis.
DS Categorized Based on Gender Distribution at Symptoms Onset | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Annually diagnosed DS participants will be categorized based on gender distribution at symptoms onset.
LGS Categorized Based on Gender Distribution at Symptoms Onset According to Stricter and Wider Diagnoses Criteria | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Annually diagnosed LGS participants will be categorized based on gender distribution at symptoms onset.
DS Categorized Based on Age Distribution at Symptoms Onset | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Annually diagnosed DS participants will be categorized based on age distribution at symptoms onset.
LGS Categorized Based on Age Distribution at Symptoms Onset According to Stricter and Wider Diagnoses Criteria | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Annually diagnosed LGS participants will be categorized based on age distribution at symptoms onset.
Diagnosis Delay for Participants With DS | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Diagnosis delay is defined as time from symptoms onset to diagnosis.
Diagnosis Delay for Participants With LGS Based on Stricter and Wider Diagnoses Criteria | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Diagnosis delay is defined as time from tonic seizures onset to electroencephalography (EEG) confirmation.
Participants With DS: Ratio of Participants Genetically and Clinically Diagnosed Versus Participants Clinically Diagnosed Only | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Participants with DS: ratio of participants genetically (Sodium Channel Protein Type 1 Subunit Alpha [SCN1A] Mutation) and clinically diagnosed versus participants clinically diagnosed only will be assessed.
Participants With LGS: Number of Participants Distributed According to Aetiologies Based on Stricter and Wider Diagnoses Criteria | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Participants with LGS: number of participants distributed according to aetiologies based on Stricter and Wider Diagnoses Criteria will be assessed.
Participants With DS: Number of Participants With Different Types of Comorbidities at Diagnosis | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Participants with DS: number of participants with different types of comorbidities at diagnosis will be assessed.
Participants With LGS: Number of Participants With Different Types of Comorbidities at Diagnosis Based on Stricter and Wider Diagnoses Criteria | At two different 12 months periods (in consecutive years at Months 12 and 24)
  Number of participants with different types of comorbidities at diagnosis based on Stricter and Wider Diagnoses Criteria will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/6b50cd656dd048fc??page=1&idFilter=TAK-935-5004